CLINICAL TRIAL: NCT04581369
Title: Cirrhosis Medical Home
Acronym: CMH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Eric Orman, Assistant Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: CMH 2003678667; R03DK122230 (NIH)
Record Dates: First submitted 2020-09-22; First posted 2020-10-09 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: Block randomization will be utilized to ensure balancing of treatment groups throughout enrollment. 20 participants will be assigned to the direct home interventions group and 20 will be assigned to standard of care.
  Caregivers (40) belong to a single arm of the study with no randomization. All receive the same study procedures.
Who Masked: Participant, Care Provider, Investigator
Masking Description: One member of the study team will randomize the participants and all other study personnel will remain blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Direct Intervention (Active Comparator): Initial Evaluation: Prior to discharge, the care coordinator will review the hospital discharge plan, obtain the approval of the patient's physicians to co-manage the patient's care, and schedule a visit with the patient at their place of discharge.
  Participants in this arm will receive direct interaction with a care coordinator to develop an individualized care plan. Frequent assessments, at least once every two weeks, will occur to continue to follow or to modify the care plan based on the needs of the patient.
  At the end of 6 months, all patients will be transitioned to receive full care by their primary care and specialty physicians and their participation in this study will be ended.
  Interventions: Other: Care Coordinator Intervention for Direct Intervention Group
- Standard of Care (Sham Comparator): Prior to hospital discharge, the care coordinator will identify the primary care and/or hepatology provider of patients in the usual care group and will ensure follow up appointments at the time of hospital discharge. The coordinator will compose and send a letter to the primary care and/or hepatology provider summarizing the patient's diagnosis, hospital course, discharge medications, and the plan of follow-up care. If the patient does not already have a primary care or hepatology provider, the coordinator will work with the patient to identify a new provider. Subjects in this group will receive no further intervention.
  Interventions: Other: Care Coordinator Intervention for Standard of Care Group
- Caregiver (Placebo Comparator): The caregivers of people with cirrhosis will be enrolled in the study. They will complete the assessments at baseline, 3 months and 6 months.
  Interventions: Other: Caregiver Intervention

INTERVENTIONS:
Other: Care Coordinator Intervention for Direct Intervention Group — The First Visit: The care coordinator will conduct a visit within 72 hours of hospital discharge to assess the patient's physical, cognitive, and psychological status, and will complete a needs assessment for both the patient and family caregiver. These measures will be used to guide the use of care protocols and development of the individualized care plan. The care plan will be developed with an emphasis on coordinating services with the patient's providers.
  The Second Visit: During the second visit, the coordinator will review the individualized care plan with both the patient and the family caregiver and will make revisions to the plan based on assessment outcomes.
  The 6-month Interaction Period: Approximately every 2 weeks, the coordinator will meet with the participant to revisit the care plan and to facilitate care.
  At the end of 6 months, all patients will be transitioned to receive full care by their primary care and specialty physicians.
  Other Names: Direct Intervention Group
  Arms: Direct Intervention
Other: Care Coordinator Intervention for Standard of Care Group — For participants randomized to this arm, a consultation with the care team will be arranged prior to hospital discharge. Outcome measures will be obtained by blinded research staff from all enrolled subjects at baseline, 3 months, and 6 months. This is the extent of interventions received for participants in this arm.
  Other Names: Standard of Care Group
  Arms: Standard of Care
Other: Caregiver Intervention — Caregivers of the participants will be assessed for caregiver burden at 3 time points.
  Arms: Caregiver

SUMMARY:
To address the health care system's lack of care coordination, the Institute of Medicine and Centers for Medicare and Medicaid Services recommend the development of collaborative care models (CCM) in a wide range of clinical settings. CCMs are intended to provide coordinated, personalized care pragmatically using care coordinators. CCMs have successfully improved care in multiple patient populations, ranging from frail older adults to depression. In contrast, for patients with cirrhosis, there is a paucity of data to support the benefit of CCM in this medically complex and vulnerable population. At Indiana University, researchers have over 20 years of experience in developing, testing, and implementing CCMs successfully for patients living with dementia or depression. Building on these successes, we have customized the CCM to best meet the unique and complex biopsychosocial needs of patients with cirrhosis: the Cirrhosis Medical Home.

DETAILED DESCRIPTION:
In the Cirrhosis Medical Home, a care coordinator, supported by an interdisciplinary clinical team, will deliver a personalized intervention guided by a set of innovative tools: (i) patient-centered care protocols, (ii) a mobile office, (iii) care coordination support software, and (iv) dynamic feedback measures.

The overall goal is to improve quality of life of patients discharged from the hospital with cirrhosis and to reduce acute health care utilization for patients with cirrhosis.

Additionally, up to 40 caregivers will be enrolled in the trial.

ELIGIBILITY:
Inclusion Criteria for patients:

* Age ≥18 years
* Cirrhosis based on:

  * biopsy
  * characteristic clinical, laboratory, and imaging findings
* Decompensated cirrhosis as denoted by either:

  * active ascites requiring paracentesis during hospitalization or
  * active overt hepatic encephalopathy requiring lactulose during hospitalization
* Poor quality of life as defined by:

  * SF-36 Physical and/or Mental Component Summary scale <40 (1SD below the mean of healthy subjects)
* Discharged to home, skilled nursing facility, sub-acute rehabilitation care, or long-term acute care
* Able to be consented, either in person or through legally authorized representative
* Access to a telephone

Inclusion criteria for caregivers:

* Age ≥18 years
* Identified caregiver of patient
* Able to be consented, either in person or through legally authorized representative
* Access to a telephone

Exclusion Criteria for patients:

* Solid organ transplant of any organ
* Life expectancy of less than 6 months
* Anticipated liver transplant within 6 months
* History of dementing illnesses and other neurodegenerative diseases such as Alzheimer's disease, Parkinson's disease, or vascular dementia
* Unable to complete study questionnaire due to hearing loss
* Legally blind
* Pregnant or nursing
* Incarcerated
* Concurrent enrollment in a related interventional research study

Exclusion criteria for caregivers:

* Impaired cognitive function
* Unable to complete study questionnaire due to hearing loss
* Legally blind
* Incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Orman, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Division of Gastroenterolgy and Hepatology, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol allowed for up to 40 caregivers to enroll in this trial. We enrolled 4 caregivers. The protocol called for 40 participants with liver disease to be enrolled and we enrolled 40. Total enrollment is 44.
Groups:
- Direct Intervention: Initial Evaluation: Prior to discharge, the care coordinator will review the hospital discharge plan, obtain the approval of the patient's physicians to co-manage the patient's care, and schedule a visit at the place of discharge.
  Participants receive direct interaction with a care coordinator to develop an individualized care plan. Frequent assessments will occur to continue to follow or to modify the care plan based on the needs of the patient.
  At the end of 6 months, all patients will be transitioned to full care by their primary care and specialty physicians and their participation in this study will be ended.
  Care Coordinator Intervention for Direct Intervention Group: The coordinator will conduct a visit within 72 hours of discharge to assess the physical, cognitive, and psychological status, and will complete a needs assessment for both the patient and family caregiver. These will be used to guide the care protocols and development of the individualized care plan. The care plan is developed with an emphasis on coordinating services with the patient's providers.
  During the second visit, the individualized care plan is reviewed with the patient and family caregiver and revisions are made based on assessment outcomes.
  The 6-month Interaction Period: The coordinator and participant meet to revisit the care plan and to facilitate care. At the end of 6 months, all patients are transitioned to full care by their primary care and specialty physicians.
Period: Overall Study
Arm/Group | Direct Intervention | Standard of Care | Caregiver
Started | 20 | 20 | 4
Completed | 4 | 4 | 4
Not Completed | 16 | 16 | 0
Not completed — Death | 7 | 6 | 0
Not completed — Lost to Follow-up | 7 | 3 | 0
Not completed — liver transplant | 2 | 2 | 0
Not completed — transitioned to hospice care | 0 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Direct Intervention | Standard of Care | Caregiver | Total
Number analyzed (Participants) | 20 | 20 | 4 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 3 | 32
  >=65 years | 6 | 5 | 1 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 2 | 29
  Male | 8 | 5 | 2 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 4 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 19 | 19 | 4 | 42
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 4 | 44

OUTCOME MEASURES:

1. Primary Outcome: Enrollment Rate
Description: The proportion of screened patients eligible, approached and enrolled will be calculated. This is an internal assessment relating not to participants but to department specific metrics.
Time Frame: Time of Enrollment
Population: Participants were screened prior to being approached for enrollment. Only after informed consent was obtained were participants randomized to a group. The numbers reported are in the aggregate for those with liver disease only and not for a particular group. Data for caregivers were not tracked.
Measure: Count of Participants; unit: Participants
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 67 | 67
Participants | 20 | 20

2. Primary Outcome: Number of Participants Who Dropped Out or Are Lost to Follow-up
Description: This is the proportion of enrolled participants (patients) who drop out of the study before completion. This is an internal assessment relating not to participants but to department specific metrics.
Time Frame: At drop out date or lost to follow-up date, which every comes first an average of 6 months
Population: Data for caregivers was not tracked. Of note we had no participants withdraw but a number were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 20 | 20
Participants | 3 | 7

3. Primary Outcome: Number of Participants With Complete Data
Description: Completeness of the data collection for enrolled subjects and reasons for incomplete data will be recorded. This is an internal assessment relating not to participants but to department specific metrics.
Time Frame: Through study completion, an average of 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Direct Intervention | Standard of Care | Caregiver
Number analyzed (Participants) | 20 | 20 | 4
Participants | 4 | 4 | 4

4. Secondary Outcome: Acute Health Care Utilization
Description: This is an assessment of patient use of health care resources, including hospitalizations and Emergency room visits. For the patient only, data will be gathered from the patient and medical record relating to the participant's emergency room visits and hospital admissions/inpatient stays during the course of their enrollment in the study.
Time Frame: 6 months
Population: Information not measured for caregivers in this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Direct Intervention | Standard of Care | Caregiver
Number analyzed (Participants) | 20 | 20 | 0
Participants | 17 | 18 | 0

5. Secondary Outcome: Health Related Quality of Life: Medical Outcome Study Short Form (SF-36)
Description: Assessment from the patient only through data collection from the Medical Outcome Study Short Form (SF-36) instrument. This 36 item questionnaire has a minimum score of 36 with a maximum score of 180; a higher score generally correlates to poorer health. This assessment was for patients only and not for caregivers.
Time Frame: measure was completed at enrollment by patients only
Population: scores at initial enrollment for patients only; caregivers were not included in this measure
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 20 | 20
score on a scale | 56 (0.7) | 58 (0.7)

6. Secondary Outcome: Health Related Quality of Life: Medical Outcome Study Short Form (SF-36)
Description: as for outcome 5
Time Frame: measure was completed at 3 months by patients only
Population: scores at 3 month enrollment for patients only; caregivers were not included in this measure
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 6 | 6
score on a scale | 84 (0.8) | 88 (0.4)

7. Secondary Outcome: Health Related Quality of Life: Medical Outcome Study Short Form (SF-36)
Description: as for outcome 5
Time Frame: measure was completed at 6 months by patients only
Population: scores at 6 month enrollment for patients only; caregivers were not included in this measure
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 4 | 4
score on a scale | 102 (0.5) | 100 (0.7)

8. Secondary Outcome: Depression Symptoms
Description: Assessment from patient only through data collection from the Patient Health Questionnaire-9 (PHQ-9) instrument. This 9 item instrument that assesses depression and has a minimum score of 0 and a maximum score of 27; a lower score generally indicates no or a lesser amount of depression/anxiety than a higher score.
Time Frame: measure was completed at initial enrollment by patients only
Population: scores at initial enrollment by patients only; caregivers were not included in this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 20 | 20
score on a scale | 11 (0.044) | 14 (0.11)

9. Secondary Outcome: Depression Symptoms
Description: as for outcome 8
Time Frame: measure was completed at 3 months by patients only
Population: scores at 3 months by patients only; caregivers were not included in this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 12 | 12
score on a scale | 14 (0.15) | 14 (0.11)

10. Secondary Outcome: Depression Symptoms
Description: as for outcome 8
Time Frame: measure was completed at 6 months by patients only
Population: scores at 6 months by patients only; caregivers were not included in this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 4 | 4
score on a scale | 12 (0.2) | 18 (0.18)

11. Secondary Outcome: Physical Performance
Description: Assessment from the patient only through data collection from the Short Physical Performance Battery (SPPB) instrument.
Time Frame: measure was completed at initial enrollment by patients only
Population: measurement was not administered so no outcome data are available
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Physical Performance
Description: Assessment from the patient only through data collection from the Short Physical Performance Battery (SPPB) instrument.
Time Frame: measure was completed at 3 months by patients only
Population: measurement was not administered so no outcome data are available
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Physical Performance
Description: Assessment from the patient only through data collection from the Short Physical Performance Battery (SPPB) instrument.
Time Frame: measure was completed at 6 months by patients only
Population: measurement was not administered so no outcome data are available
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Anxiety Symptoms
Description: Assessment from patient only through data collection from the Generalized Anxiety Disorder Scale (GAD-7) instrument. This 7 item instrument that assess anxiety has a minimum score of 0 and a maximum score of 21, with a lower score indicating no or lesser anxiety than a higher score.
Time Frame: measure was completed at initial enrollment by patients only
Population: scores at initial enrollment by patients only; caregivers were not included in this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 9 | 12
units on a scale | 7 (0.11) | 9 (0.11)

15. Secondary Outcome: Anxiety Symptoms
Description: as for outcome 14
Time Frame: measure was completed at 3 months by patients only
Population: scores at 3 months by patients only; caregivers were not included in this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 7 | 18
units on a scale | 14 (0.11) | 14 (0.15)

16. Secondary Outcome: Anxiety Symptoms
Description: as for outcome 14
Time Frame: measure was completed at 6 months by patients only
Population: scores at 6 months by patients only; caregivers were not included in this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 12 | 18
units on a scale | 16 (0.2) | 16 (0.2)

17. Secondary Outcome: Cognitive Assessment With 3D CAM (Confusion Assessment Method)
Description: Assessment of overall levels of cognitive status, including hepatic encephalopathy
Time Frame: measure was completed at initial enrollment by patients only
Population: measurement was not administered so no outcome data are available
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Cognitive Assessment With 3D CAM (Confusion Assessment Method)
Description: Assessment of overall levels of cognitive status, including hepatic encephalopathy
Time Frame: measure was completed at 3 months by patients only
Population: measurement was not administered so no outcome data are available
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Cognitive Assessment With 3D CAM (Confusion Assessment Method)
Description: Assessment of overall levels of cognitive status, including hepatic encephalopathy
Time Frame: measure was completed at 6 months by patients only
Population: measurement was not administered so no outcome data are available
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Cognitive Assessment With PHES (The Psychometric Hepatic Encephalopathy Score)
Description: Assessment of overall levels of cognitive status, including hepatic encephalopathy. PHES range is -18 to +6. Normal is > -4 (better). <= -5 is abnormal (worse).
Time Frame: measure was completed at initial enrollment by patients only
Population: scores at initial enrollment by patients only; caregivers were not included in this measure
Measure: Count of Participants; unit: Participants
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 18 | 17
Participants
  score >-5 | 7 | 3
  score ≤-5 | 11 | 14

21. Secondary Outcome: Cognitive Assessment With PHES (The Psychometric Hepatic Encephalopathy Score)
Description: as for outcome 20
Time Frame: measure was completed at 3 month enrollment by patients only
Population: scores at 3 month enrollment by patients only; caregivers were not included in this measure
Measure: Count of Participants; unit: Participants
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 3 | 4
Participants
  score >-5 | 3 | 3
  score ≤-5 | 0 | 1

22. Secondary Outcome: Cognitive Assessment With PHES (The Psychometric Hepatic Encephalopathy Score)
Description: as for outcome 20
Time Frame: measure was completed at 6 month enrollment by patients only
Population: scores at 6 month enrollment by patients only; caregivers were not included in this measure
Measure: Count of Participants; unit: Participants
Arm/Group | Direct Intervention | Standard of Care
Number analyzed (Participants) | 2 | 2
Participants
  score >-5 | 2 | 1
  score ≤-5 | 0 | 1

23. Secondary Outcome: Caregiver Burden
Description: Assessment from caregivers only through data collection from the Zarit Burden Interview-12 (ZBI-12) instrument; a lower score is generally indicative of a lower amount caregiver fatigue or perception of burden; a higher score generally correlates to a greater level of caregiver fatigue/perceived burden.
  0-10 no burden, 10-20 mild-moderate burden, >20 high burden. Minimum: 0 Maximum: 48
Time Frame: caregivers completed at initial enrollment--while the plan was to complete at 3 and 6 months, none of the participants with liver disease for whom these people cared were alive at the 3 and 6 month mark so the instruments were not completed
Population: Caregivers of patients with liver disease who enrolled in the Cirrhosis Medical Home study were eligible for study enrollment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Caregivers: Caregivers of patients with liver disease who enrolled in the Cirrhosis Medical Home study were eligible for study participation as well. Caregiver participation involved completion of the Zarit 12 caregiver burden survey
Arm/Group | Caregivers
Number analyzed (Participants) | 4
units on a scale | 10 (0.5)

ADVERSE EVENTS:
Time Frame: 6 months
Description: We utilized the same verbiage to classify adverse events, both regular and serious as found in the clincialtrials.gov definitions.
Arm/Group | Direct Intervention | Standard of Care | Caregiver
All-Cause Mortality (participants affected / at risk) | 7/20 | 6/20 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/4
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT04581369/Prot_SAP_000.pdf